CLINICAL TRIAL: NCT02996942
Title: Key Aspects of Medical Practice in Patients With Haemophilia A
Acronym: KAPPA
Status: Withdrawn | Type: Observational
Why Stopped: Not active
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/118
Record Dates: First submitted 2014-05-19; First posted 2016-12-19 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Joint Disease
Keywords: haemophilia, joint disease, quality of life
MeSH Terms: conditions — Joint Diseases; Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Replacement therapy: Hemophilia A receiving replacement therapy (prophylaxis or on demand)
  Interventions: Biological: Factor VIII replacement

INTERVENTIONS:
Biological: Factor VIII replacement — Patients receive their usual treatment
  Other Names: factor VIII

SUMMARY:
The KAPPa project has the aim to create an international database in which information about clinical features, therapeutic management, burden of illness and costs of severe and moderate haemophilia A patients from different countries and sites is collected. The aim of this project is to analyse the influence of such different characteristics on medical, psychosocial and economic outcomes in patients over the long-term.

DETAILED DESCRIPTION:
1000 patients with hemophilia A will be enrolled using a webbased registry. Key quality factors that will be registered are : hemophilia joint Health score (HJHS), annual bleed rate, quality of Life (EQ5D), as well as dosing of replacement therapy.

ELIGIBILITY:
Inclusion Criteria: or forms.

* severe haemophilia A (factor VIII<1%)
* moderate (factor VIII<5%)
* signed informed consent

Exclusion Criteria:

* Not fullfilling inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from haemophilia centers.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Outcome of factor replacement treatment | 3 years
  Joint disase according to HJHS. Quality of Life. Health economic evalaution.

IPD SHARING:
Plan to Share IPD: Undecided